CLINICAL TRIAL: NCT02203266
Title: A Randomised, Parallel-group, Multi-centre Trial Using a Novel INCA Tracker Device to Measure and Monitor Compliance and Technique of Seretide Diskus Inhaler in a Community Pharmacy Setting
Brief Title: Teaching Inhaler Use With the INCA Device in a Community Pharmacy Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beaumont Hospital (Other)
Collaborators: Royal College of Surgeons, Ireland (Other)
Responsible Party: Principal Investigator, Professor Richard Costello, Professor Richard Costello, Beaumont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC004
Record Dates: First submitted 2014-07-27; First posted 2014-07-29 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Asthma; Pulmonary Disease, Chronic Obstructive
Keywords: Medication Adherence; Patient Compliance
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive; Medication Adherence; Patient Compliance | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Feedback (Experimental): Feedback on the patient's own inhaler use, with personalized information on the patients technique and timing of use of the diskus inhaler as recorded on the INCA device will be provided to patients in the feedback group after 1,2 and 6 months.
  Interventions: Device: Feedback
- Demonstration (Active Comparator): Current best practice - inhaler technique education
  Interventions: Behavioral: Education
- Control (No Intervention): Usual care in the community pharmacy setting

INTERVENTIONS:
Device: Feedback — Feedback on the patient's own inhaler use, with personalized information on the patients technique and timing of use of the diskus inhaler as recorded on the INCA device will be provided to patients in the feedback group after 1,2 and 6 months.
  Other Names: INCA Device
  Arms: Feedback
Behavioral: Education — Feedback on the patient's own inhaler technique as observed by pharmacist and education to support best use will be provided to patients in the demonstration group after 1,2 and 6 months.
  Arms: Demonstration

SUMMARY:
The purpose of this trial is to discover whether providing feedback to patients from a device that records when and how well a patient uses a Seretide Diskus inhaler will lead to:

* Improved compliance with prescribed inhaler use
* Improved technique of inhaler use
* A reduction in respiratory health related outcomes caused by poor inhaler compliance and usage.
* An improvement in patient quality of life scores

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years old or above
* Capable of understanding and willing to provide voluntary informed consent before any protocol specific procedures are performed
* Capable of understanding and complying with the requirements of the protocol, and demonstrating a willingness to attend for all required visits.
* Able and willing to take inhaled medication.
* Have a valid prescription for use of a Seretide diskus inhaler or already using a Seretide diskus inhaler.
* Have a history of regular attendance in the pharmacy in which they are recruited which will be demonstrated by the subject having collected three prescriptions for any medication in that pharmacy in the six months preceeding their recruitment to the study.

Exclusion Criteria:

* Patient expressly reports that their physician has indicated that they will not be continuing to receive Seretide over the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2014-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Rate of adherence | 2 months and 6 months
  The rate of adherence is the proportion of correctly taken drugs at the correct time relative to the prescribed interval.

SECONDARY OUTCOMES:
Rescue inhaled medication use | Six months
Rescue antibiotic and/or steroid medication use | 6 months
Quality of life | 2 months and 6 months
Adherence in the time domain | Two months and six months
Technique adherence | Two months and six months

CONTACTS AND LOCATIONS:
Overall Officials: Richard Costello, Professor, Principal Investigator — Royal College of Surgeons in Ireland, Clinical Research Centre, Beaumont Hospital
Locations (1):
- Boots Retail (Ireland) Limited, Dublin, Ireland

REFERENCES:
- [Derived] O'Dwyer SM, MacHale E, Sulaiman I, Holmes M, Hughes C, D'Arcy S, Rapcan V, Taylor T, Boland F, Bosnic-Anticevich S, Reilly RB, Ryder SA, Costello RW. The effect of providing feedback on inhaler technique and adherence from an electronic audio recording device, INCA(R), in a community pharmacy setting: study protocol for a randomised controlled trial. Trials. 2016 May 4;17(1):226. doi: 10.1186/s13063-016-1362-9. PMID 27142873